CLINICAL TRIAL: NCT06881251
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo- and Active-controlled, Dose Ranging Study to Evaluate the Efficacy and Safety of JNJ-95475939 for the Treatment of Participants With Moderate to Severe AD
Brief Title: A Study of JNJ-95475939 in the Treatment of Participants With Moderate to Severe Atopic Dermatitis (AD)
Acronym: DUPLEX-AD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 95475939ADM2001; 95475939ADM2001 (Other: Janssen Research & Development, LLC); 2024-517814-13-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A: Dupilumab (Active Comparator): Participants will receive Dupilumab dose regimen 1 subcutaneously through Week 22.
  Interventions: Drug: Dupilumab
- Group B: JNJ-95475939 (Experimental): Participants will receive JNJ-95475939 dose regimen 1 subcutaneously through Week 22.
  Interventions: Drug: JNJ-95475939
- Group C: JNJ-95475939 (Experimental): Participants will receive JNJ-95475939 dose regimen 2 subcutaneously through Week 22.
  Interventions: Drug: JNJ-95475939
- Group D: JNJ-95475939 (Experimental): Participants will receive JNJ-95475939 dose regimen 3 subcutaneously through Week 22.
  Interventions: Drug: JNJ-95475939
- Group E: Placebo (Placebo Comparator): Participants will receive matching placebo subcutaneously through Week 10, then switch to receive JNJ-95475939 dose regimen 1 subcutaneously between Week 12 and Week 22.
  Interventions: Drug: JNJ-95475939; Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Dupilumab will be administered subcutaneously.
  Arms: Group A: Dupilumab
Drug: JNJ-95475939 — JNJ-95475939 will be administered subcutaneously.
  Arms: Group B: JNJ-95475939; Group C: JNJ-95475939; Group D: JNJ-95475939; Group E: Placebo
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Group E: Placebo

SUMMARY:
The purpose of this study is to evaluate how well JNJ-95475939 works as compared to placebo in participants with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion criteria:

* Chronic Atopic Dermatitis (AD), according to American Academy of Dermatology Consensus Criteria with onset of symptoms at least 1 year prior to the screening visit
* Eczema Area and Severity Index (EASI) score greater than and equal to (>=) 16 at the screening and baseline visits
* Validated investigator global assessment for AD (vIGA-AD) score >= 3 at the screening and baseline visits
* >= 10% body surface area (BSA) of AD involvement at the screening and baseline visits
* Baseline Peak Pruritus Numeric(al) Rating Scale (PP-NRS) average score of >=4
* Documented history (within 6 months before screening) of either inadequate response or inadvisability to topical treatments, or inadequate response to systemic therapies (within 12 months before screening)
* Participant has applied a moisturizer at least once daily for at least 7 days before the baseline visit

Exclusion criteria:

* Experienced primary efficacy failure (no response within 16 weeks) or an adverse event (AE) requiring discontinuation related to agents (eg, severe ocular surface disease, dupilumab-associated facial redness) inhibiting IL-4Rα, IL-4, and/or IL-13 signaling (eg, dupilumab, lebrikizumab, or tralokinumab)
* Participant is pregnant or breastfeeding, or planning to become pregnant or breastfeed during the study
* Active skin disease other than AD including eczema herpeticum, molluscum contagiosum, impetigo, psoriasis or has any other ongoing significant skin condition including skin infections, that, according to the investigator, could interfere with efficacy assessments
* Current diagnosis or signs or symptoms of severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Recent case of eczema herpeticum, herpes zoster within 8 weeks before screening, or history of recurrent eczema herpeticum
* History of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (eg, untreated latent tuberculosis), recurrent urinary tract infection, fungal infection, mycobacterial infection, or open, draining, or infected skin wounds, or ulcers.
* Diagnosed active parasitic infection or at high risk of parasitic infection, unless treated with antihelminth therapy prior to randomization
* Had major surgery (eg, requiring general anesthesia and hospitalization), within 8 weeks before screening, or will not have fully recovered from surgery, or has such surgery planned during the time the participant is expected to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Eczema Area and Severity Index (EASI) 75 Response at Week 12 | Baseline, Week 12
  EASI-75 response is defined as at least 75 percent (%) improvement in EASI total score. EASI-75 response is defined as at least 75% improvement from baseline in EASI total score. The EASI score is used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.

SECONDARY OUTCOMES:
Percentage of Participants With EASI-90 Response at Week 12 | Baseline, Week 12
  EASI-90 response is defined as at least 90% improvement in EASI total score. EASI-90 response is defined as at least 90% improvement from baseline in EASI total score. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants With EASI-100 Response at Week 12 | Baseline, Week 12
  EASI-100 response is defined as at least 100% improvement in EASI total score. EASI-100 response is defined as at least 100% improvement from baseline in EASI total score. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Score of 0 or 1 and a Reduction From Baseline of Greater Than Equal to (>=) 2 Points at Week 12 | Baseline, Week 12
  vIGA-AD is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0, where 0=Clear: No inflammatory signs of AD; 1=almost clear: Barely perceptible erythema, induration/papulation and/or lichenification; 2=mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting; 3=moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present and 4=severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present. Higher scores are indicative of a more severe AD.
Percentage of Participants Achieving vIGA-AD Score of 0 and a Reduction From Baseline of >= 2 Points at Week 12 | Baseline, Week 12
  vIGA-AD is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0, where 0=Clear: No inflammatory signs of AD; 1=almost clear: Barely perceptible erythema, induration/papulation and/or lichenification; 2=mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting; 3=moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present and 4=severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present. Higher scores are indicative of a more severe AD.
Percent Change From Baseline in the EASI Total Score at Week 12 | Baseline, Week 12
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants Achieving a >= 4-Point Reduction in Skin Pain Numerical Rating Scale (NRS) Score From Baseline to Week 12 | Baseline, Week 12
  The Skin Pain NRS is a single item asking participants to assess their worst skin pain over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change from Baseline in Peak Pruritus Numerical Rating Scale (PP-NRS) Score at Week 12 | Baseline, Week 12
  The PP-NRS is a single item asking participants to assess their worst itch over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change from Baseline in Skin Pain NRS Score at Week 12 | Baseline, Week 12
  The Skin Pain NRS is a single item asking participants to assess their worst skin pain over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change from Baseline in the Score of Item 2 of the AD Sleep Scale at Week 12 | Baseline, Week 12
  The AD sleep scale is a validated 3-item PRO instrument to capture self-reported impact of itch on sleep disturbance each day, including difficulty falling asleep, number of night-time awakenings, and difficulty falling back asleep after waking during the previous night. Each AD Sleep Scale item is scored individually. For Item 2, participants select the number of times they woke up each night, ranging from 0 to 29 times.
Percentage of Participants Achieving a >= 4-Point Reduction in PP-NRS Score From Baseline Through Week 12 | From Baseline through Week 12
  The PP-NRS is a single item asking participants to assess their worst itch over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percentage of Participants with EASI-75 Response at Week 16 | Baseline, Week 16
  EASI-75 response is defined as at least 75% improvement in EASI total score. EASI-75 response is defined as at least 75% improvement from baseline in EASI total score. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants with EASI-90 Response at Week 16 | Baseline, Week 16
  EASI-90 response is defined as at least 90% improvement in EASI total score. EASI-90 response is defined as at least 90% improvement from baseline in EASI total score. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants with EASI-100 Response at Week 16 | Week 16
  EASI-100 response is defined as at least 100% improvement in EASI total score. EASI-100 response is defined as at least 100% improvement from baseline in EASI total score. The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants Achieving vIGA-AD Score of 0 or 1 and a Reduction From Baseline of >= 2 Points at Week 16 | Baseline, Week 16
  vIGA-AD is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0, where 0=Clear: No inflammatory signs of AD; 1=almost clear: Barely perceptible erythema, induration/papulation and/or lichenification; 2=mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting; 3=moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present and 4=severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present. Higher scores are indicative of a more severe AD.
Percentage of Participants Achieving vIGA-AD Score of 0 and a Reduction From Baseline of >= 2 Points at Week 16 | Baseline, Week 16
  vIGA-AD is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0, where 0=Clear: No inflammatory signs of AD; 1=almost clear: Barely perceptible erythema, induration/papulation and/or lichenification; 2=mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting; 3=moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present and 4=severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present. Higher scores are indicative of a more severe AD.
Percent Change from Baseline in the EASI Total Score at Week 16 | Baseline, Week 16
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants Achieving a >= 4-Point Reduction in Skin Pain Numerical Rating Scale (NRS) Score From Baseline to Week 16 | Baseline, Week 16
  The Skin Pain NRS is a single item asking participants to assess their worst skin pain over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change from Baseline in PP-NRS Score at Week 16 | Baseline, Week 16
  The PP-NRS is a single item asking participants to assess their worst itch over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change from Baseline in Skin Pain NRS Score at Week 16 | Baseline, Week 16
  The Skin Pain NRS is a single item asking participants to assess their worst skin pain over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change from Baseline in the Score of Item 2 of the AD Sleep Scale at Week 16 | Baseline, Week 16
  The AD sleep scale is a validated 3-item PRO instrument to capture self-reported impact of itch on sleep disturbance each day, including difficulty falling asleep, number of night-time awakenings, and difficulty falling back asleep after waking during the previous night. Each AD Sleep Scale item is scored individually. For Item 2, participants select the number of times they woke up each night, ranging from 0 to 29 times.
Percentage of Participants Achieving a >= 4-Point Reduction in PP-NRS Score From Baseline Through Week 24 | From Baseline Through Week 24
  The PP-NRS is a single item asking participants to assess their worst itch over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percentage of Participants with EASI-75 Response at Week 24 | Baseline, Week 24
  EASI-75 response is defined as at least 75% improvement in EASI total score. EASI-75 response is defined as at least 75% improvement from baseline in EASI total score. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants with EASI-90 Response at Week 24 | Week 24
  EASI-90 response is defined as at least 90% improvement in EASI total score. EASI-90 response is defined as at least 90% improvement from baseline in EASI total score. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants with EASI-100 Response at Week 24 | Week 24
  EASI-100 response is defined as at least 100% improvement in EASI total score. EASI-100 response is defined as at least 100% improvement from baseline in EASI total score. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants Achieving vIGA-AD Score of 0 or 1 and a Reduction From Baseline of >= 2 Points at Week 24 | Baseline, Week 24
  vIGA-AD is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0, where 0=Clear: No inflammatory signs of AD; 1=almost clear: Barely perceptible erythema, induration/papulation and/or lichenification; 2=mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting; 3=moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present and 4=severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present. Higher scores are indicative of a more severe AD.
Percentage of Participants Achieving vIGA-AD Score of 0 and a Reduction From Baseline of >= 2 Points at Week 24 | Baseline, Week 24
  vIGA-AD is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0, where 0=Clear: No inflammatory signs of AD; 1=almost clear: Barely perceptible erythema, induration/papulation and/or lichenification; 2=mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting; 3=moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present and 4=severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present. Higher scores are indicative of a more severe AD.
Percent Change from Baseline in the EASI Total Score at Week 24 | Baseline, Week 24
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting a higher severity of AD.
Percentage of Participants Achieving a >= 4-Point Reduction in Skin Pain NRS Score From Baseline to Week 24 | Baseline, Week 24
  The Skin Pain NRS is a single item asking participants to assess their worst skin pain over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change From Baseline in PP-NRS Score at Week 24 | Baseline, Week 24
  The PP-NRS is a single item asking participants to assess their worst itch over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change from Baseline in Skin Pain NRS Score at Week 24 | Baseline, Week 24
  The Skin Pain NRS is a single item asking participants to assess their worst skin pain over the past 24 hours. The response categories range from 0 (no pain) to 10 (worst pain). Higher scores indicating greater severity.
Percent Change from Baseline in the Score of Item 2 of the AD Sleep Scale at Week 24 | Baseline, Week 24
  The AD sleep scale is a validated 3-item PRO instrument to capture self-reported impact of itch on sleep disturbance each day, including difficulty falling asleep, number of night-time awakenings, and difficulty falling back asleep after waking during the previous night. Each AD Sleep Scale item is scored individually. For Item 2, participants select the number of times they woke up each night, ranging from 0 to 29 times.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Baseline up to Week 36
  Participants with AEs and SAEs will be reported. An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product. TEAEs are AEs with onset during the intervention phase or that are a consequence of a preexisting condition that has worsened since baseline. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Locations (71):
- United States (13):
  - First OC Dermatology, Fountain Valley, California
  - University of California Los Angeles - Division of Dermatology, Los Angeles, California
  - Hamilton Research LLC, Alpharetta, Georgia
  - DeNova Research, Chicago, Illinois
  - Dawes Fretzin Clinical Research Group LLC, Indianapolis, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Red River Research Partners LLC, Fargo, North Dakota
  - Optima Research, Boardman, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - Arlington Center for Dermatology, Arlington, Texas
  - Center for Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Frontier Derm Partners CRO, LLC, Mill Creek, Washington
- Argentina (4):
  - CIPREC, Buenos Aires
  - INAER - Investigación en Alergias y Enfermedades Respiratorias, Buenos Aires
  - Instituto de Neumonologia y Dermatologia, Buenos Aires
  - Derma Internacional S A, Buenos Aires
- Brazil (6):
  - Ceti - Centro de Estudos Em Terapias Inovadoras, Curitiba
  - Hospital De Clinicas De Porto Alegre, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Fundacao do ABC Centro Universitario FMABC, Santo André
  - BR TRIALS Ensaios Clinicos e Consultoria Ltda, São Paulo
- Canada (7):
  - Dermatology Research Institute Inc, Calgary, Alberta
  - Dr. Chih ho Hong Medical, Surrey, British Columbia
  - Karma Clinical Trials Inc., St. John's, Newfoundland and Labrador
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre De Recherche Dermatologique Du Quebec Metropolitain, Québec, Quebec
- Germany (9):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite - Universitaetsmedizin Berlin (CCM), Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Hautarztpraxis, Bramsche
  - Medizinische Fakultaet Carl Gustav Carus Technische Universitaet Dresden, Dresden
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Universitatsklinikum Frankfurt, Frankfurt
  - Eurofins bioskin GmbH, Hamburg
  - Studienzentrum Dr Schwarz Germany, Langenau
- Japan (10):
  - Fukuoka University Hospital, Fukuoka
  - Osaka Habikino Medical Center, Habikino
  - Teikyo University Hospital, Itabashi Ku
  - Kume Clinic, Sakai
  - Sapporo Skin Clinic, Sapporo
  - Jitaikai Tachikawa dermatology clinic, Tachikawa
  - Shirasaki Dermatology Clinic, Takaoka Shi
  - Mie University Hospital, Tsu
  - Queens Square Medical Facilities, Yokohama
  - Nomura Dermatology Clinic, Yokohama
- Poland (10):
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Care Clinic, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Centrum Medyczne All Med, Krakow
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno Badawczy Marek Brzewski Pawel Brzewski Spolka Cywilna, Krakow
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - Therapia Nova, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - WroMedica I Bielicka A Strzalkowska s c, Wroclaw
- Spain (7):
  - Hosp. Gral. Univ. Dr. Balmis, Alicante
  - Hosp. Univ. San Cecilio, Granada
  - Hosp. Univ. de Bellvitge, LHospitalet de Llobregat
  - Grupo Dermatologico Y Estetico Pedro Jaen, Madrid
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. de Manises, Manises
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
- United Kingdom (5):
  - The Queen Elizabeth Hospital King's Lynn NHS Foundation Trust, Kings Lynn
  - Royal London Hospital, London
  - Northwick Park Hospital, London
  - Guys and St Thomas NHS Foundation Trust, London
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency